CLINICAL TRIAL: NCT04461535
Title: Corticotropin Stimulation in Adrenal Venous Sampling for Patients With Primary Aldosteronism The ADOPA Randomized Clinical Trial
Brief Title: Corticotropin Stimulation in Adrenal Venous Sampling for Patients With Primary Aldosteronism(ADOPA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor.Qifu Li, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ADOPA study
Record Dates: First submitted 2020-06-22; First posted 2020-07-08 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; adrenal venous sampling; adrenocorticotropic hormone
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVS with ACTH stimulation (Experimental): Patients divided into AVS with ACTH stimulation group need to undergo stimulation with a continuous cosyntropin infusion.
  Interventions: Drug: Adrenocorticotropic hormone
- AVS without ACTH stimulation (No Intervention): Patients divided into AVS without ACTH stimulation group take the same procedure of AVS with a continuous saline infusion.

INTERVENTIONS:
Drug: Adrenocorticotropic hormone — Patients divided into Intervention group need to undergo stimulation with a continuous cosyntropin infusion (50 μg/h started 30 minutes before sampling during AVS). Right and left adrenal venous blood and corresponding peripheral venous blood should be sampled sequentially.
  Other Names: ACTH
  Arms: AVS with ACTH stimulation

SUMMARY:
To compare the effect of different procedures of AVS(with or without ACTH stimulation) on the long-term outcomes of patients with PA

DETAILED DESCRIPTION:
This is a prospective and randomized study involving patients with primary aldosteronism(PA) who completed AVS.

All paticipants will be randomized into ACTH-stimulated group(Intervention group) and ACTH-unstimulated group(Control group) Cannulation was considered successful when the selectivity index (SI), namely plasma cortisol concentration (PCC) in adrenal vein/PCC in IVC≥3 with ACTH stimulation or SI≥2 without ACTH stimulation. The ratio of PAC: PCC on the side with the higher ratio over the contralateral PAC: PCC ratio is defined as the lateralization index (LI). Lateralization of aldosterone excess was defined as LI≥4 irrespective of ACTH use. Patients with LI between 2 and 4 together with contralateral suppression (PAC/PCC of non-dominant side < PAC/PCC of IVC) or CT showing a typical adenoma on the dominant side were also considered to have lateralized disease. Patients with LI < 2 or LI 2-4 without meeting the above criteria were diagnosed as BPA.

In case of technical AVS failure or bilateral PAC/PCC in adrenal venous blood lower than peripheral blood, if the patient meets one of the following criteria, adrenalectomy was recommended: 1) unilateral nodule on CT (≥ 1 cm), no observable nodules or hyperplasia on contralateral adrenal, and PAC ≥ 20 ng/dl, PRC < 5 μIU/ml, K ≤ 3.5mmol/l; 2) unilateral nodule on CT (≥ 1 cm), no observable nodules or hyperplasia on contralateral adrenal, and the contralateral index≤0.5 in AVS.

Surgical intervention is recommended for unilateral PA (UPA) whereas bilateral PA (BPA) is typically treated with oral mineralocorticoid receptor antagonists such as spironolactone. The aim is to compare the long-term outcomes of patients with PA.

To evaluate whether the treatment decision (surgical or medical treatment) based on different AVS procedures (with or without ACTH stimulation) would lead to different outcomes in patients with PA.

ELIGIBILITY:
1.Inclusion criteria: Patients who meet the following criterion can be included in this study.

1. Aged between 18-70, male or female, with legal capacity
2. PA diagnosis confirmed by at least one confirmatory test: positive PA screening (ARR≥ 2.0 ng·dl-1/IU·l-1) and at least one positive PA confirmatory test (PAC-post CCT ≥11 ng/dl, PAC-post SSIT≥8·0 ng/dl, or if confirmatory tests were in grey zone (i.e, PAC 8-11 ng/ml two hours after administration of 50 mg captopril or PAC 60-80 pg/ml after the infusion of 2L normal saline), PAC-post FST≥6·0 ng/dl);

2.Exclusion criteria: Patients with one of the following conditions will be excluded in this study:

1. refusal by the patient to undergo AVS or adrenalectomy;
2. meeting the criteria for bypassing AVS [i.e. younger than 35 years old, with typical aldosterone-producing adenomas characteristics (plasma aldosterone >30ng/dl, serum potassium <3·5mmol/l, CT indicated unilateral 1cm low-density adenoma) ;
3. allergic to ACTH or contrast media;
4. pregnant or lactating women;
5. patients with a history of uncontrolled malignant tumor;
6. complicated with Cushing's syndrome [including subclinical Cushing: cortisol after 1mg dexamethasone suppression test (DST)>138 nmol/l or cortisol after 1mg DST 50-138 nmol/l plus adrenocorticotrophic hormone (ACTH)<10pg/ml;
7. diagnosed with familial hyperaldosteronism;
8. with imaging characteristics suggestive of pheochromocytoma or adrenal cortical carcinoma;
9. patients unsuitable for surgery, such as those with heart failure (New York Heart Association (NYHA) class III or IV), severe anemia (Hemoglobin<60g/L), stroke or acute coronary syndrome within 3 months, severe ascites and cirrhosis, estimated glomerulus filtration rate<30ml/min/m2;
10. with alcohol or drug abuse and active mental health disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of surgically treated patients with complete biochemical remission in the overall cohort between two groups | At 12 months of follow-up.
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
Compare the proportion of surgically treated patients who achieved complete clinical remission in the overall cohort between two groups | At 12 months of follow-up.
  The proportion of complete clinical remission according to PASO consensus criteria.Clinical outcomes were determined by the blood pressure response to treatment and the number and dosage of antihypertensive medications.
Daily defined doses (DDD) of antihypertensive agents (including MRA), blood pressure, proportion of patients reaching target blood pressure | At 12 months of follow-up.
  Daily defined doses (DDD) of antihypertensive agents (including MRA), blood pressure, proportion of patients reaching target blood pressure in each group irrespective of their treatment after 12 months of follow-up
Rate of bilaterally successful AVS | At baseline.
  Calculate the rate of bilateral successful catheterization.Successful catheterization was defined as SI≥2 without ACTH stimulation or SI≥3 with ACTH stimulation.
Adverse events | At baseline and 12 month of follow-up.
  Record the occurrence of adverse events, including adrenal venous hemorrhage and related adrenal insufficiency, hypertensive urgencies, anaphylactic shock, venous thrombosis, pulmonary embolism, ect.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Nishikawa T, Omura M, Satoh F, Shibata H, Takahashi K, Tamura N, Tanabe A; Task Force Committee on Primary Aldosteronism, The Japan Endocrine Society. Guidelines for the diagnosis and treatment of primary aldosteronism--the Japan Endocrine Society 2009. Endocr J. 2011;58(9):711-21. doi: 10.1507/endocrj.ej11-0133. Epub 2011 Aug 9. PMID 21828936
- [Result] Deinum J, Groenewoud H, van der Wilt GJ, Lenzini L, Rossi GP. Adrenal venous sampling: cosyntropin stimulation or not? Eur J Endocrinol. 2019 Sep;181(3):D15-D26. doi: 10.1530/EJE-18-0844. PMID 31176302
- [Result] Buffolo F, Monticone S, Williams TA, Rossato D, Burrello J, Tetti M, Veglio F, Mulatero P. Subtype Diagnosis of Primary Aldosteronism: Is Adrenal Vein Sampling Always Necessary? Int J Mol Sci. 2017 Apr 17;18(4):848. doi: 10.3390/ijms18040848. PMID 28420172
- [Result] Dekkers T, Prejbisz A, Kool LJS, Groenewoud HJMM, Velema M, Spiering W, Kolodziejczyk-Kruk S, Arntz M, Kadziela J, Langenhuijsen JF, Kerstens MN, van den Meiracker AH, van den Born BJ, Sweep FCGJ, Hermus ARMM, Januszewicz A, Ligthart-Naber AF, Makai P, van der Wilt GJ, Lenders JWM, Deinum J; SPARTACUS Investigators. Adrenal vein sampling versus CT scan to determine treatment in primary aldosteronism: an outcome-based randomised diagnostic trial. Lancet Diabetes Endocrinol. 2016 Sep;4(9):739-746. doi: 10.1016/S2213-8587(16)30100-0. Epub 2016 Jun 17. PMID 27325147
- [Result] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Derived] Yang S, Du Z, Zhang X, Zhen Q, Shu X, Yang J, Song Y, Yang Y, Li Q, Hu J; Chongqing Primary Aldosteronism Study (CONPASS) Group. Corticotropin Stimulation in Adrenal Venous Sampling for Patients With Primary Aldosteronism: The ADOPA Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2338209. doi: 10.1001/jamanetworkopen.2023.38209. PMID 37870836